CLINICAL TRIAL: NCT00926003
Title: Neuropsychological Benefits of Cognitive Training in Ugandan HIV Children
Brief Title: Computerized Cognitive Rehabilitation in Ugandan Children With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Global Health Uganda LTD (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Michael J. Boivin, Professor of Psychiatry and Neurology & Ophthalmology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIRB 07-709; R34MH085631 (Other Grant/Funding Number: National Institute of Health)
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: HIV Infections
Keywords: HIV; Children; Africa; Neuropsychology; cognitive rehabilitation; computers
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full Computerized Cognitive Training (Experimental): Intervention is a Computer Cognitive Rehabilitation Training delivered in 24 sessions over 8 weeks (3 times/week). A training session lasts about an hour and consists of 9 training games or programs, 3 pertaining to improving attention, 3 pertaining to improving visual-spatial memory, and 3 pertaining to improving reasoning/planning. Each training game become more difficult as the child gains proficiency.
  Interventions: Behavioral: Full Computerized cognitive training
- Control (No Intervention): Passive Control with no intervention training (computer cognitive games) for 8 weeks.
- Limited computerized cognitive training (Active Comparator): Intervention is a Computer Cognitive Rehabilitation Training delivered in 24 sessions over 8 weeks (3 times/week). A training session lasts about an hour and consists of 9 training games or programs, 3 pertaining to improving attention, 3 pertaining to improving visual-spatial memory, and 3 pertaining to improving reasoning/planning. In this arm, however, the training games do NOT become progressively more difficult as the child gains proficiency, but rotates randomly among simpler to moderate levels of difficulty for each game. The purpose to to give children int he "limited" CCRT arm comparable exposure to the cognitive games training as with the "full CCRT" arm, with the exception of the titrating nature of the game training.
  Interventions: Behavioral: Limited computerized cognitive training

INTERVENTIONS:
Behavioral: Full Computerized cognitive training — 8 weeks of 3 times weekly intervention for 60 min per session with the full titrating version of Captain's Log program (3 games for attention, 3 games for visual spatial working memory, 3 games for reasoning/planning
  Other Names: computerized cognitive games; computerized cognitive rehabilitation therapy (CCRT)
  Arms: Full Computerized Cognitive Training
Behavioral: Limited computerized cognitive training — Locked Captain's Log CCRT that rotates randomly among simplest level of computer cognitive games training. 8 weeks of 3 times weekly intervention for 60 min per session with the non-titrating version of Captain's Log program (3 games for attention, 3 games for visual spatial working memory, 3 games for reasoning/planning).
  Other Names: computerized cognitive rehabilitation therapy (CCRT)
  Arms: Limited computerized cognitive training

SUMMARY:
One-hundred and fifty-nine school-age children with HIV in Kayunga District, Uganda were randomized to one of 3 treatment arms: 24 training sessions of a computerized cognitive rehabilitation therapy (CCRT) program called Captain's Log; 24 sessions of Captain's Log not titrated to child's performance; or no training intervention. Study Aim 1: To compare the neuropsychological benefit of 24 training sessions of Captain's Log CCRT to the active and passive control groups over a 8-week period, and at 3-month follow-up. Study Aim 2: To compare the psychiatric benefit of 24 training sessions of Captain's Log CCRT to the active and passive control groups over an 8-week period, and at 3-month follow-up. Study Aim 3: To evaluate how ART treatment status, and the corresponding clinical stability of the child modifies CCRT neuropsychological performance gains and psychiatric symptom reduction. Outcome Assessments: The Kaufman Assessment Battery for Children, 2nd ed. (KABC-2), Tests of Variables of Attention (TOVA) visual and auditory tests, CogState computerized neuropsychological screening test, Bruininks-Oseretsky Test of Motor Proficiency (BOT-2), and Achenbach Child Behavior Checklist (CBCL) will be administered before and after the 8-week training period and at 3-month follow-up post training. Captain's Log has an internal evaluator feature which will help us monitor the specific training tasks to which the children best respond. Analyses: We will compare neuropsychological and psychiatric gains over the 8-week training period and at 3-mo follow-up for our three study groups, anticipating that they will be significantly greater for the CCRT intervention children (Study Aims 1 & 2). These neuropsychological gains will be associated with improved school performance over the long-term. Intervention children clinically stable on ART will have greater gains than those not stable or virally suppressed on ART. Conclusion: CCRT will prove effective and sustainable for enhancing neurocognitive status in HIV children. Futher work will prove this approach viable for assessing and treating children in resource-poor settings.

DETAILED DESCRIPTION:
Aim 1. To evaluate the effectiveness of CCRT in improving cognitive performance outcomes in Ugandan children with HIV.

Hypothesis 1a: CCRT can improve short and long-term cognitive outcomes in children with HIV; Hypothesis 1b: Improvements in performance associated with CCRT are not solely due to increased computer exposure.

One-hundred and fifty school-age children with HIV in Kayunga District, Uganda, will undergo baseline neuropsychological testing using the Kaufman Assessment Battery for Children (KABC-2), the computerized Tests of Variables of Attention (TOVA: auditory and visual tests), the brief CogState computerized neuropsychological test battery (CogState), and the Bruininks-Oseretsky Tests of Motor Proficiency (2nd edition) (BOT-2). Cogstate is designed as a neuropsychological screening tool with minimal practice effects and suitable in a repeated measures design for monitoring the benefits of treatment on neurocognitive disability11. Children then will be randomized to either: CCRT intervention group (Captain's Log active rehabilitation), active control group (Captain's Log locked, non-rehabilitation mode), or passive control group (no computer intervention). CCRT or computer controls will be presented over 24 sessions (~ 45 min) for 8 weeks (3 sessions per week). After the 8-weeks, neurocognitive gains will be assessed with CogState and the KABC-2 working memory subscales (primary expected outcome measures). The full KABC-2, TOVA, CogState, and BOT-2 will be re-administered 3 months after the 8-week assessment. Thus, the full battery will be administered at enrollment and at 3-month follow-up, while the most strategic portions of the battery will be administered following the 8 weeks CCRT intervention period. The combined testing will allow us to assess both the short-term and longer-term neuropsychological benefits of CCRT.

Aim 2. To evaluate the effectiveness of CCRT in reducing psychiatric symptoms in Ugandan children with HIV.

Hypothesis 2: CCRT can reduce short- and long-term psychiatric symptoms in children with HIV.

Previously in cerebral malaria survivors, we demonstrated a significant reduction in short-term symptoms related to anxiety, depression, and somatic complaints as assessed by the Achenbach Child Behavior Checklist (CBCL) following CCRT intervention12. In this aim, caregiver-reported psychiatric symptoms on the CBCL will be assessed at enrollment, after the 8-week CCRT intervention period, and 3 months after enrollment. The CBCL assessment will also help us gauge the psychosocial benefits of the social attention and enrichment surrounding computer exposure in the active control condition, rather than the rehabilitative aspects of CCRT per se. This will be evident as we compare the active and passive control groups.

Aim 3. To evaluate how ARV treatment status and clinical response along with corresponding immunological status of the child modifies CCRT neuropsychological performance gains and psychiatric symptom reduction; .after controlling for quality of home environment, nutrition, and other risk factors of poverty.

Hypothesis 3: Children virally suppressed on ART treatment with a history of fewer opportunistic illnesses and better CD4 counts will have better neuropsychological outcomes in response to CCRT training.The moderating effects of HIV progressive encephalopathy on brain plasticity can also be monitored by CCRT training progress, measures by the Captain's Log Internal Evaluator (CLIE) feature of the CCRT program.

ELIGIBILITY:
Inclusion Criteria:

* HIV children 6 to 16 years of age and enrolled in the CAI program will be eligible should the parent or caregiver consent to participation in the study. They will all be confirmed HIV positive children (ELISA and Western blot). Only children with perinatally acquired HIV infection will be included.

Exclusion Criteria:

* At pre-CCRT medical examination (see medical exam form in appendices) we will exclude children with a medical history of serious birth complications, severe malnutrition, bacterial meningitis, encephalitis, cerebral malaria, or other known brain injury or disorder requiring hospitalization. Also children with seizure or other neurological disability will be excluded. This will be screened using a brief medical history questionnaire and CAI medical chart review.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Boivin, PhD, MPH, Study Director — MSU Psychiatry
Locations (1):
- Global Health Uganda, Kampala, Uganda

REFERENCES:
- [Result] Ruisenor-Escudero H, Familiar I, Nakasujja N, Bangirana P, Opoka R, Giordani B, Boivin M. Immunological correlates of behavioral problems in school-aged children living with HIV in Kayunga, Uganda. Glob Ment Health (Camb). 2015 Jun 25;2:e9. doi: 10.1017/gmh.2015.7. eCollection 2015. PMID 28596857
- [Result] Giordani B, Novak B, Sikorskii A, Bangirana P, Nakasujja N, Winn BM, Boivin MJ. Designing and evaluating Brain Powered Games for cognitive training and rehabilitation in at-risk African children. Glob Ment Health (Camb). 2015 May 29;2:e6. doi: 10.1017/gmh.2015.5. eCollection 2015. PMID 28596854
- [Result] Boivin MJ, Nakasujja N, Sikorskii A, Opoka RO, Giordani B. A Randomized Controlled Trial to Evaluate if Computerized Cognitive Rehabilitation Improves Neurocognition in Ugandan Children with HIV. AIDS Res Hum Retroviruses. 2016 Aug;32(8):743-55. doi: 10.1089/AID.2016.0026. Epub 2016 May 2. PMID 27045714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 159 school-age clinically stable children receiving monthly out-patient care at the Walter Reed Children's Clinic at the Kayunga District Hospital Kayunga town, Uganda.
Pre-assignment Details: Of 190 total available children at the study site, 159 were enrolled into the present clinical trial. 13 were ineligible due to profound neurocognitive disability or very poor health; 7 could not be reached; 7 lived outside of the study catchment area, and 4 declined to participate.
Groups:
- CCRT Intervention: Computer Cognitive Rehabilitation Training Intervention 24 sessions over 8 weeks
  Computerized cognitive rehabilitation therapy (CCRT): 8 weeks of 3 times weekly intervention for 45 min per session with Captain's Log program
- Control: Passive Control with no intervention training for 8 weeks
- Limited CCRT: Locked CCRT that does not become more difficult with mastery of child on computer games training
  Limited CCRT active control intervention: Locked Captain's Log CCRT that rotates randomly among simplest level of computer cognitive games training
Period: Baseline
Arm/Group | CCRT Intervention | Control | Limited CCRT
Started | 53 | 54 | 52
Completed | 53 | 54 | 52
Not Completed | 0 | 0 | 0
Period: Post-Training Evaluation
Arm/Group | CCRT Intervention | Control | Limited CCRT
Started | 53 | 54 | 52
Completed | 52 | 54 | 52
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Post-Training 3-month Follow-up
Arm/Group | CCRT Intervention | Control | Limited CCRT
Started | 52 | 54 | 52
Completed | 51 | 54 | 52
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCRT Intervention | Control | Limited CCRT | Total
Number analyzed (Participants) | 53 | 54 | 52 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.7) | 8.8 (1.9) | 8.7 (2.0) | 8.9 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 30 | 81
  Male | 29 | 27 | 22 | 78

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Performance (KABC2)
Description: Kaufman Assessment Battery for Children, 2nd edition (KABC-II) Mental Processing Index (MPI), which is a global cognitive ability performance composite that is a standard score with a mean of 100 and a standard deviation of 15, with scores for our population of children typically ranging from 55 to 130. the MPI is comprised of the standardized global scores for the cognitive domains of Sequential Processing, Simultaneous Processing, Learning, and Planning. These standardized global domain scores are summed and converted (on the basis of age of child, using American norms) to a composite global performance measure called the Mental Processing Index (MPI) standard score (T score). Higher T scores indicate better performance and a better neuropsychological outcome.
Time Frame: KABC-II MPI score at post-training 3 mo follow-up assessment, adjusted for baseline KABC-II MPI performance. Therefore, only a single score appears in the table.
Measure: Mean (Standard Error); unit: T scores from USA norms for this test
Arm/Group | CCRT Intervention | Control | Limited CCRT
Number analyzed (Participants) | 53 | 54 | 52
T scores from USA norms for this test | 63.32 (0.60) | 61.13 (0.57) | 62.65 (0.62)
Statistical Analysis 1: Comparison: CCRT Intervention vs Control vs Limited CCRT; Least Square Means from Longitudinal Model, Their Standard Errors by Trial Arm Adjusted for Age, Being on ART at Intake, Socioeconomic Score, Home Score, Recruitment Location, KABC Learning and Delayed Recall Scores at Baseline, and Outcome Score at Baseline; Test type: Superiority; p = 0.02, ANCOVA

2. Secondary Outcome: Achenbach Child Behavior Checklist (CBCL) Total Score
Description: Child Behavior Checklist (CBCL) total score Total problems T-scores (standardized). This is a standardized score with a mean of 50 and a standard deviation of 10, with higher scores indicating more symptoms of either emotional (internalizing) or behavioral (externalizing) or other (e.g., sleep disturbances) nature. Range for our children on this scale is typically from 40 to 80. These are t scores based on Cross-Cultural norms, whereby higher scores (more symptoms or problems) indicate a worse outcome.
Time Frame: CBCL total score at post-training (3 months), adjusted by the baseline score, so that a single score appears in the results table.
Population: 3-mo follow-up means adjusted for outcome at baseline, ARV treatment status
Measure: Mean (Standard Error); unit: T scores based on cross cultural norms
Arm/Group | CCRT Intervention | Control | Limited CCRT
Number analyzed (Participants) | 51 | 54 | 52
T scores based on cross cultural norms | 55.61 (0.83) | 54.45 (0.78) | 53.46 (0.86)
Statistical Analysis 1: Comparison: CCRT Intervention vs Control vs Limited CCRT; Least Square Means from Longitudinal Model, Their Standard Errors by Trial Arm Adjusted for Age, Being on ARV at Intake, Socioeconomic Score, Home Score, Recruitment Location, KABC Learning and Delayed Recall Scores at Baseline, and Outcome Score at Baseline; Test type: Superiority; p = 0.18, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were in surveillance during entire study time period
Groups:
- CCRT Intervention: Intervention is a Computer Cognitive Rehabilitation Training delivered in 24 sessions over 8 weeks (3 times/week)
  Computerized cognitive rehabilitation therapy (CCRT): 8 weeks of 3 times weekly intervention for 45 min per session with Captain's Log program
Arm/Group | CCRT Intervention | Control | Limited CCRT
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 0/51 | 0/54 | 0/52

LIMITATIONS AND CAVEATS:
Uganda Ministry of Health mandated ARV treatment of all children with HIV part way through the trial. Future research should replicate our findings using CCRT with children with HIV already stabilized on ARV treatment and virally supporessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No